CLINICAL TRIAL: NCT03276039
Title: Serum Pentraxin-3 in Non-alcoholic Fatty Liver Disease With or Without Hepatitis C Virus: A Comparative Egyptian Study
Brief Title: Serum Pentraxin-3 in Non-alcoholic Fatty Liver Disease With or Without Hepatitis C Virus
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shereen Abou Bakr Saleh, Assistant Professor, Ain Shams University
Other Study IDs: 456
Record Dates: First submitted 2017-09-02; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 25 patients with non-alcoholic fatty liver disease
  Interventions: Diagnostic Test: plasma pentraxin-3
- 25 patients with NAFLD and chronic HCV
  Interventions: Diagnostic Test: plasma pentraxin-3
- 20 healthy controls
  Interventions: Diagnostic Test: plasma pentraxin-3

INTERVENTIONS:
Diagnostic Test: plasma pentraxin-3 — Plasma pentraxin-3 was measured using ELISA

SUMMARY:
This study included 70 subjects divided into 3 groups. Group I included 25 patients with NAFLD. Group II included 25 patients with NAFLD and chronic HCV. Group III: included 20 controls. Abdominal ultrasound was done to patients and controls. Plasma pentraxin-3 (PTX3) was measured using ELISA. Comparison between three groups was done regarding plasma pentraxin-3. Higher levels of plasma PTX3 were detected in NAFLD patients irrespective of presence or absence of chronic HCV infection. Plasma PTX3 could be used as a non-invasive test for prediction of metabolic syndrome in the high-risk population with high sensitivity and moderate specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NAFLD.
* Patients with NAFLD and chronic hepatitis C viral infection.

Exclusion Criteria:

* Current or past consumption of significant amount of alcohol more than 21 drinks and 14 drinks per week for men and women respectively.
* Patients receiving Drugs which cause fatty liver as amiodarone, diliazem, tamoxifen, steroids.
* Patients who take statins as it has lowering effect on plasma PTX3.
* Patients having any clinical evidence of hepatic decompensation, such as hepatic encephalopathy, ascites, variceal bleeding, elevated serum bilirubin level to more than two folds the upper limit of normal.
* Patients with heart failure.
* Patients with autoimmune rheumatic disease.
* Patients with chronic kidney diseases.
* Patients with sepsis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 adult Egyptian patients collected from Gastroenterology Unit, Internal Medicine, and Tropical Medicine Departments, were included. Additionally, 20 apparently healthy subjects were included as the control group. They were classified into three groups: Group I: included 25 patients with NAFLD diagnosed by radiological features and by exclusion of other causes of fatty liver.
  Group II: included 25 patients with radiological features of NAFLD and laboratory evidence of chronic hepatitis C viral infection (positive PCR).
  Group III: included 20 apparently healthy control subjects with negative medical history, normal physical examination, and normal laboratory and radiological examination.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Plasma pentraxin-3 as a non invasive diagnostic marker in diagnosis of NAFLD in comparison to it's levels in patients with NAFLD and chronic hepatitis C viral infection | 1 year
  Measurement of plasma pentraxin-3 in patients with NAFLD in comparison to it's levels in patients with hepatic steatosis on top of HCV and normal controls